CLINICAL TRIAL: NCT03006289
Title: Relationship of Metabolic Syndrome and Its Components With Thyroid Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Lin Liao (Other)
Responsible Party: Sponsor-Investigator, Lin Liao, chief of endocrinology department at Qianfoshan Hospital, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: qfsnfm-003
Record Dates: First submitted 2016-12-26; First posted 2016-12-30 (Estimated); Last update posted 2016-12-30 (Estimated); Status verified 2016-12

CONDITIONS: Thyroid Cancer
Keywords: Metabolic Syndrome; fasting plasma glucose
MeSH Terms: conditions — Thyroid Neoplasms; Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- The thyroid cancer group: The postoperative pathology of thyroid is malignant
- The thyroid nodule group: The postoperative pathology of thyroid is benign

SUMMARY:
The purpose of this study is to investigate the association between metabolic syndrome (MS), body mass index (BMI), hyperglycemia, dyslipidemia, hypertension and thyroid cancer. Screen for the risk factors that affect the incidence of thyroid cancer.

ELIGIBILITY:
Inclusion Criteria:

1. patients undergone thyroid surgery
2. signed the informed consent

Exclusion Criteria:

1.patients with no surgery

Ages: 8 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients undergone thyroid surgery
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-10 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
lipids | before the thyroid surgery

SECONDARY OUTCOMES:
glucose | before the thyroid surgery

OTHER OUTCOMES:
blood pressure | before the thyroid surgery
Uric Acid | before the thyroid surgery
sialic acid | before the thyroid surgery
thyroid function | before the thyroid surgery

CONTACTS AND LOCATIONS:
Overall Officials: Lin Liao, MD, Study Chair — Qianfoshan Hospital

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Yao J, Zhao J, Liu J, Jiang S, Guo S, Xu L, Zhang X, Sheng Q, Wang K, Liao L, Dong J. The relationships between thyroid functions of short-term rapid hypothyroidism and blood lipid levels in post-thyroidectomy patients of differentiated thyroid cancer. Front Endocrinol (Lausanne). 2023 Apr 27;14:1114344. doi: 10.3389/fendo.2023.1114344. eCollection 2023. PMID 37181036
- [Derived] Zhao J, Tian Y, Jia Z, Yao J, Liao L, Dong J. Abnormal Glucose Metabolism Parameters and the Aggressiveness of Differentiated Thyroid Carcinoma: A Hospital-Based Cross-Section Study in China. Front Endocrinol (Lausanne). 2022 Mar 1;13:806349. doi: 10.3389/fendo.2022.806349. eCollection 2022. PMID 35299970
- [Derived] Zhao J, Tian Y, Yao J, Gu H, Zhang R, Wang H, Liao L, Dong J. Hypercholesterolemia Is an Associated Factor for Risk of Differentiated Thyroid Cancer in Chinese Population. Front Oncol. 2021 Jan 28;10:508126. doi: 10.3389/fonc.2020.508126. eCollection 2020. PMID 33585179